CLINICAL TRIAL: NCT03764592
Title: Mapping of Ventricular Fibrillation (VF) Substrates and VF Arrhythmogenic Sources/Reentrant Circuits in Patients With Brugada and Early Repolarization Syndromes
Brief Title: VF Mapping in Brugada and Early Repolarization Syndromes
Status: Completed | Type: Observational
Sponsor: Pacific Rim Electrophysiology Research Institute (Other)
Collaborators: University of Bordeaux (Other)
Responsible Party: Principal Investigator, Koonlawee Nademanee, MD, Principal Investigator, Pacific Rim Electrophysiology Research Institute
Other Study IDs: PACIFICReri2
Record Dates: First submitted 2018-12-03; First posted 2018-12-05 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Brugada Syndrome; Early Repolarization Syndrome
MeSH Terms: conditions — Brugada Syndrome | interventions — Radiofrequency Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- VF BrS/ERS patients: Only patients that diagnosed with BrS or ERS based on ECG criteria
  Interventions: Other: radiofrequency ablation

INTERVENTIONS:
Other: radiofrequency ablation — Symptomatic patients whose substrates were identified will undergo catheter ablation; asymptomatic patients will be followed without undergoing catheter ablation.

SUMMARY:
To determine the values and limitations of ECGI in guiding ablation and risk stratification in patients with BrS and Early Repolarization.

DETAILED DESCRIPTION:
The investigators will study symptomatic BrS and ERs syndrome (N=25) and asymptomatic patients (N=25) age between 16-70 years old to determine values and limitations of non-invasive mapping using electrocardiographic imaging (ECGI) in identifying VF substrates as target sites for catheter ablations in patients with Brugada (BrS) and Early repolarization syndromes (ERS) and also determine the mechanisms of VF in BrS and ERs syndromes.

ELIGIBILITY:
Inclusion Criteria:

Patients presenting with the type1 BrS ECG or ER ECG signature pattern, with/without a sodium channel blocker. Patients with the following one of these symptoms or arrhythmias will be considered as symptomatic patients: 1) aborted cardiac arrest cases, 2) documented VF episodes, 3) agonal respiration during sleep with difficulty to arouse, 4) syncope of unknown origin, or 5) seizure suspected of arrhythmic origin.•

Exclusion Criteria:

Patients who refuse informed consent and to participate to the best ability in the study.

Patients who have structural heart disease or concomitant medical illness.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Brugada marker or early repolarization marker on ECG.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-02-23 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
VF death | 3 years
  ventricular fibrillation

CONTACTS AND LOCATIONS:
Overall Officials: Koonlawee Nademanee, MD, Principal Investigator — Chulalongkorn University
Locations (2):
- Thailand (2):
  - Bumrungrad International Hospital, Bangkok
  - Pacific Rim Electrophysiology Research Institute Data Coordinating Center, Bangkok

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nademanee K, Raju H, de Noronha SV, Papadakis M, Robinson L, Rothery S, Makita N, Kowase S, Boonmee N, Vitayakritsirikul V, Ratanarapee S, Sharma S, van der Wal AC, Christiansen M, Tan HL, Wilde AA, Nogami A, Sheppard MN, Veerakul G, Behr ER. Fibrosis, Connexin-43, and Conduction Abnormalities in the Brugada Syndrome. J Am Coll Cardiol. 2015 Nov 3;66(18):1976-1986. doi: 10.1016/j.jacc.2015.08.862. PMID 26516000
- [Result] Nademanee K, Hocini M, Haissaguerre M. Epicardial substrate ablation for Brugada syndrome. Heart Rhythm. 2017 Mar;14(3):457-461. doi: 10.1016/j.hrthm.2016.12.001. Epub 2016 Dec 12. No abstract available. PMID 27979714
- [Result] Nademanee K, Veerakul G, Chandanamattha P, Chaothawee L, Ariyachaipanich A, Jirasirirojanakorn K, Likittanasombat K, Bhuripanyo K, Ngarmukos T. Prevention of ventricular fibrillation episodes in Brugada syndrome by catheter ablation over the anterior right ventricular outflow tract epicardium. Circulation. 2011 Mar 29;123(12):1270-9. doi: 10.1161/CIRCULATIONAHA.110.972612. Epub 2011 Mar 14. PMID 21403098
- [Result] Veerakul G, Nademanee K. Will we be able to cure brugada syndrome? Heart Rhythm. 2016 Nov;13(11):2159-2160. doi: 10.1016/j.hrthm.2016.08.025. Epub 2016 Aug 17. No abstract available. PMID 27544747